CLINICAL TRIAL: NCT06742359
Title: Relationship of Magnetic Resonance Imaging Parameters with Shoulder Function and Pain in Patients with Subacromial Impingement Syndrome
Brief Title: Magnetic Resonance Imaging Parameters in Patients with Subacromial Impingement Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24/455
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial impingement syndrome; pain; function; magnetic resonance imaging
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with subacromial impingement syndrome

SUMMARY:
Shoulder pain is the third most common musculoskeletal pain complaint in the world with an incidence of 7-30%. Subacromial impingement syndrome (SIS) is the most common cause of shoulder pain. Imaging in impingement syndrome is usually based on different imaging modalities. X-ray, magnetic resonance imaging (MRI) and ultrasound are the most commonly used, and MRI is considered by many authors to be the most reliable imaging modality for evaluation of the rotator cuff because it allows evaluation of soft tissues as well as bony abnormalities such as subacromial osteophytes and acromioclavicular joint capsular hypertrophy. MRI allows the diagnosis of rotator cuff tears with greater interobserver reliability than ultrasound in assessing tear size, retraction and atrophy. Few studies have investigated the impact of pathologic findings on MRI on the degree of symptoms and functional impairment seen in these patients. The aim of this study was to investigate the relationship between shoulder pain and function and MRI findings in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
In this clinical study, 100 patients who were admitted to Fatih Sultan Mehmet Training and Research Hospital Physical Medicine and Rehabilitation outpatient clinic with shoulder pain and diagnosed with subacromial shoulder impingement by routine laboratory and imaging tests will be included in this study. Demographic data such as age, gender, body mass index, education, occupation, comorbidities, smoking, alcohol consumption will be recorded. Pain intensity will be assessed by Visual analog scale (VAS) and function will be assessed by Shoulder Pain and Disability Index (SPADI).

Pain Assessment: The VAS is a one-dimensional measure of pain intensity and is commonly used in adult populations including rheumatologic patients. It can be used horizontally or vertically. The patient marks his/her own pain on a 10 cm ruler with no pain at one end and the most severe pain at the other end. In this method, the patient is told that there are two extremes and that he/she is free to mark any point between these points.

Functional assessment: All patients will be assessed for shoulder function using the Shoulder Pain and Disability Index (SPADI) The SPADI is a self-administered questionnaire that includes two dimensions, one for pain and one for functional activities. In the pain dimension, there are five questions about the severity of an individual's pain. Eight questions assess functional activities designed to measure the degree of difficulty an individual has in performing various activities of daily living that require the use of the upper limbs. Patients are asked to place a 10 cm mark as the answer to each question.

Shoulder joint range of motion: Participants' shoulder range of motion (ROM) active and passive flexion, abduction, internal and external rotation will be examined with a goniometer.

Magnetic resonance imaging: All MRI scans will be reviewed by an independent radiologist specializing in musculoskeletal imaging who is unaware of the patients' clinical data. Each MRI scan will include at least one transverse, sagittal and coronal plane consisting of at least one T1-weighted and at least one proton density (PD) weighted or T2-weighted fat-suppressed sequence. All MRI parameters will be electronically evaluated using a PACS workstation (SimplexBT PACS, Ankara Universitesi Teknokent, Ankara, Turkey).

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-65
2. Shoulder pain for at least six weeks

Exclusion Criteria:

1. Presence of a rheumatologic disease,
2. Presence of neurological disease
3. Pregnancy
4. Symptomatic osteoarthritis of the shoulder, shoulder instability, pathologies of the tendon of the long head of the biceps, glenoid injuries and partial tears greater than 3 mm and full-thickness tears of the rotator cuff
5. Corticosteroid, hyaluronic acid and/or PRP injection in the shoulder area within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subacromial impingement syndrome.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 2 months
  Pain Assessment: The visual analog scale is a one-dimensional measure of pain intensity and is widely used in adult populations, including rheumatologic patients. It can be used horizontally or vertically. The patient marks their pain on a 10 cm ruler with no pain at one end and the most severe pain at the other. Patients are asked to rank their pain intensity on a 10-point scale, where 0 = no pain, 5 = moderate pain and 10 = unbearable pain. In this method, the patient is told that there are two extremes and that they are free to mark any point in between. A higher value indicates more severe pain.

SECONDARY OUTCOMES:
Function | 2 months
  Functional assessment: All groups will be assessed for shoulder function using the Shoulder Pain and Disability Index. The Shoulder Pain and Disability Index includes two dimensions, one for pain and one for functional activities. Patients are asked to describe the extent of their shoulder problems by marking a number on a scale from zero (no pain or disability) to ten (maximum pain and disability) for each item. The results from each subscale are then summed and converted into a score out of 100. A minimum score of 0 and a maximum score of 100 can be obtained. The higher the final score, the greater the shoulder pain, impairment or disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No